CLINICAL TRIAL: NCT00983281
Title: Use of Hextend in Trauma
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Kenneth Proctor, Professor, University of Miami
Other Study IDs: 20080598
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Results first posted 2013-02-18 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2013-02

CONDITIONS: Trauma
Keywords: Combat casualty care; Hextend; Colloid
MeSH Terms: conditions — Wounds and Injuries | interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hextend: Patients that received Hextend as part of their fluid resuscitation.
  Interventions: Drug: Hextend
- Standard of Care: Patients that received standard fluid resuscitation but no Hextend.
  Interventions: Drug: Hextend

INTERVENTIONS:
Drug: Hextend — IV fluid resuscitation to restore euvolemia after traumatic injury and surgery.

SUMMARY:
This is a chart review of all trauma patients during the specified time period. The purpose of this study is to examine the effects of resuscitation with hextend after trauma, in the adult population. The authors hypothesize that when compared to patients resuscitated with standard of care, resuscitation with Hextend will result in a mortality difference.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the trauma center

Exclusion Criteria:

* Pregnant women, children, psychiatric patients and prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma patients
Sampling Method: Probability Sample
Enrollment: 1714 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Proctor, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Hextend: Patients that received Hextend as part of their resuscitation fluid.
- Standard of Care: Patients that received standard of care but no Hextend as part of their resuscitation.
Period: Overall Study
Arm/Group | Hextend | Standard of Care
Started | 805 | 909
Completed | 805 | 909
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hextend | Standard of Care | Total
Number analyzed (Participants) | 805 | 909 | 1714
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean Age | 39 (17) | 41 (18) | 40 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 190 | 342
  Male | 653 | 719 | 1372

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Time Frame: Overall inpatient mortality upon discharge from the hospital with a mean length of stay of 8 days.
Measure: Number; unit: participants
Groups:
- Standard of Care: PAtients that did not receive Hextend as part of their resuscitation fluid.
Arm/Group | Hextend | Standard of Care
Number analyzed (Participants) | 805 | 909
participants | 42 | 81

ADVERSE EVENTS:
Description: Serious and/or other (non-serious) adverse events were not collected or assessed as part of this observational study.
Groups:
- Standard of Care: Patients that received standard resuscitation but no Hextend as part of their resuscitation.
Arm/Group | Hextend | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No